CLINICAL TRIAL: NCT06167252
Title: Map of Unwanted Loneliness
Status: Completed | Type: Observational
Sponsor: José Joaquín Mira Solves (Other)
Collaborators: Centro Internacional para la Investigación del Envejecimiento (Unknown)
Responsible Party: Sponsor-Investigator, José Joaquín Mira Solves, Professor, Fundación para el Fomento de la Investigación Sanitaria y Biomédica de la Comunitat Valenciana
Organization: Fundación para el Fomento de la Investigación Sanitaria y Biomédica de la Comunitat Valenciana (Other)
Other Study IDs: UGP-23-189
Record Dates: First submitted 2023-12-04; First posted 2023-12-12 (Actual); Last update posted 2025-04-01 (Actual); Status verified 2025-03

CONDITIONS: Loneliness

STUDY DESIGN:
Observational Model: Ecologic or Community | Time Perspective: Retrospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Other: Exploration of a database — extraction of data

SUMMARY:
Creating a map of the magnitude of the problem and the response of primary care to unwanted loneliness among the elderly, stratifying different needs based on place of residence and proximity to available assistance programs to address this issue, which, due to its scale, calls for collaboration among various institutions, disciplines, and experiences.

ELIGIBILITY:
Inclusion Criteria:

* Population aged 65 or older.
* Registration of medical records related to unanticipated loneliness.
* Patients with diagnoses of anxiety disorders (CIE-10 F41.1, F41.2, F41.8, F41.9, F43.2, F45, F48) or insomnia (CIE-10 F51) or affective disorders (CIE-10 F34.1) or somatization (CIE-10 F45.0) or pathological grief (CIE-10 Z63.4) or those referred to mental health or social worker services.

Exclusion Criteria:

* None

Min Age: 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Older Adult
Study Population: Population aged 65 or older who attend one of the 10 primary care centers participating in the provinces of Alicante and Valencia between March 1, 2022, and December 31, 2023.
Sampling Method: Non-Probability Sample
Enrollment: 992 (Actual)
Dates: Start 2022-05-01 (Actual); Primary Completion 2023-11-30 (Actual); Study Completion 2023-12-31 (Actual)

PRIMARY OUTCOMES:
NH | 21 months
  Number of hospitalizations

SECONDARY OUTCOMES:
NFMV | 21 months
  Number of family medicine visits
NPCNV | 21 months
  Number of primary care nursing visits
NPSWV | 21 months
  Number of primary care social work visits
NFPV | 21 months
  Number of primary care physiotherapy visits
NCPHV | 21 months
  Number of primary care home consultations
NCEPV | 21 months
  Number of primary care emergency consultations
NHD | 21 months
  Number of hospitalization days
NTDMGE | 21 months
  Number of total daily medications (general and related to emotional condition)
NTEM | 21 months
  Number of total daily medications (related only to emotional condition)

CONTACTS AND LOCATIONS:
Locations (1):
- FISABIO, Alicante, Spain

IPD SHARING:
Plan to Share IPD: Undecided